CLINICAL TRIAL: NCT04097925
Title: Doravirine Concentrations and Antiviral Activity in Genital Fluids in HIV-1 Infected Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other); Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Daniel Podzamczer, Chief of the HIV and STD Unit (Infectious Disease Service), Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DORAGEN; 2018-003921-27 (EudraCT Number)
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Results first posted 2022-05-25 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: HIV-1-infection
Keywords: Doravirine
MeSH Terms: interventions — doravirine; emtricitabine tenofovir alafenamide

STUDY DESIGN:
Intervention Model Description: Patients with Doravirine administered orally once daily in combination with Tenofovir alafenamide (TAF) and emtricitabine (FTC) co-formulated as single tablet (Descovy® TAF/FTC) and administered orally once daily.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Doravirine + Descovy® TAF/FTC (Experimental): Doravirine (MK-1439) 100 mg administered orally once daily in combination with Tenofovir alafenamide (TAF) and emtricitabine (FTC) co-formulated as single tablet (Descovy® TAF/FTC 25/200 mg) and administered orally once daily during 16 weeks
  Interventions: Drug: Doravirine; Drug: Descovy

INTERVENTIONS:
Drug: Doravirine — Doravirine 100 mg tablet
  Other Names: MK-1439
Drug: Descovy — Tenofovir alafenamide 25 mg / emtricitabine 200 mg tablet
  Other Names: TAF/FTC

SUMMARY:
This study aims to evaluate the ability of Doravirine to penetrate the genital tract and suppress viral replication and provide evidence for the use of Doravirine as part of treatment strategies as prevention.

DETAILED DESCRIPTION:
Objectives:

* To determine Doravirine concentrations in seminal plasma and cervicovaginal fluid in HIV-1 infected male and female individuals receiving antiretroviral therapy (ATR) with Doravirine plus Descovy®.
* To evaluate HIV-1 viral load in seminal plasma and cervicovaginal fluid in HIV-1 infected male and female individuals receiving ART with Doravirine plus Descovy®.

Study Phase:

Phase II

Study Design:

Open label, single arm, single center, prospective study.

Study Disease:

HIV-1 infection

Study Endpoints:

* Concentration of Doravirine in seminal plasma and cervicovaginal fluid in HIV-1 infected male and female individuals, respectively, 8 weeks after switching to Doravirine plus Descovy®.
* HIV-1 RNA in seminal plasma and cervicovaginal fluid in HIV-1 infected male and female individuals, respectively, 8 weeks after switching to Doravirine plus Descovy®.

Target Population:

Male and female adult HIV-1 infected patients receiving standard ART with tenofovir alafenamide/emtricitabine (TAF/FTC), tenofovir disoproxil fumarate/emtricitabine or abacavir/lamivudine , plus an non-nucleoside reverse transcriptase inhibitor, a boosted protease inhibitor or an integrase inhibitor during at least 3 months, with plasma HIV-1 RNA suppression (<40 copies/mL) during at least 6 months.

Number of Subjects Planned:

15 male and 15 female individuals.

Study duration:

16 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Asymptomatic, HIV-1 infected individuals ≥ 18 years of age.
2. Be on a stable ART consisting of TAF/FTC, tenofovir disoproxil fumarate/emtricitabine or abacavir/lamivudine, plus an non-nucleoside reverse transcriptase inhibitor, a boosted protease inhibitor or an integrase inhibitor, continuously for at least 3 consecutive months preceding the screening visit.
3. Plasma HIV-1 RNA <40 copies/mL for at least 6 months at the Screening visit.
4. Signed and dated written informed consent prior to inclusion.
5. Female Subjects of Childbearing Potential must agree to utilize a highly effective method of contraception during heterosexual intercourse from the screening visit throughout the duration of the study.

Exclusion Criteria:

1. Severe hepatic impairment (Child-Pugh Class C)
2. Ongoing malignancy
3. Active opportunistic infection
4. Resistance to any of the antiretroviral (ARV) included in the study or history of virologic failure with risk of resistance selection to any of the study drugs.
5. Any verified Grade 4 laboratory abnormality
6. ALT or AST ≥ 3xULN and/or bilirubin ≥ 1.5xULN
7. Severe renal impairment (Estimated creatinine filtration rate <50mL/min).
8. Females who are pregnant (as confirmed by positive serum pregnancy test) or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Podzamczer Palter, PhD Chief, Principal Investigator — Hospital Universitari de Bellvitge
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Doravirine + Descovy® TAF/FTC
Started | 30
Completed | 29
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Doravirine + Descovy® TAF/FTC
Number analyzed (Participants) | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 41 [23 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Spain | 30

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Doravirine in Seminal Plasma Fluid
Description: Concentration of Doravirine in seminal plasma fluid in HIV-1 infected male individuals
Time Frame: 8 weeks after switching (from baseline visit) to Doravirine plus TAF/FTC
Population: Descriptive analysis was performed for male participants (15), defining median and IQR of Doravirine concentrations in seminal plasma
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Doravirine + Descovy® TAF/FTC
Number analyzed (Participants) | 15
ng/ml | 127 [31.2 to 272]

2. Primary Outcome: Concentration of Doravirine in Cervicovaginal Fluid
Description: Concentration of Doravirine in cervicovaginal fluid in HIV-1 infected female individuals
Time Frame: 8 weeks after switching to Doravirine plus TAF/FTC
Population: Descriptive analysis was performed for female participants (14), defining median and IQR of Doravirine concentrations in CVF
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Doravirine + Descovy® TAF/FTC
Number analyzed (Participants) | 14
ng/ml | 505.8 [199.8 to 960.8]

3. Primary Outcome: Number of Participants With HIV-1 RNA Seminal Plasma <40 Copies/mL
Description: Number of participants with HIV-1 RNA seminal plasma <40 Copies / mL of HIV measured by real-Time Reverse Transcriptase Polymerase Chain Reaction Amplification
Time Frame: 8 weeks after switching (from baseline visit) to Doravirine plus TAF/FTC
Population: Number of patients with HIV-1 RNA seminal plasma <40 copies/ml
Measure: Number; unit: Number of participants
Arm/Group | Doravirine + Descovy® TAF/FTC
Number analyzed (Participants) | 15
Number of participants | 15

4. Primary Outcome: Quantification of Participants With HIV-1 RNA <40 Copies / mL in Cervicovaginal Fluid
Description: Number of participants with HIV-1 RNA cervicovaginal fluid<40 Copies / mL of HIV measured by real-Time Reverse Transcriptase Polymerase Chain Reaction Amplification
Time Frame: 8 weeks after switching (from baseline visit) to Doravirine plus TAF/FTC
Population: Number of patients with HIV-1 RNA cervicovaginal fluid <40 copies/ml
Measure: Number; unit: Number of participants
Arm/Group | Doravirine + Descovy® TAF/FTC
Number analyzed (Participants) | 15
Number of participants | 14

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Doravirine + Descovy® TAF/FTC
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 18/30
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doravirine + Descovy® TAF/FTC (N=30)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Trichomonas vaginal infection (Infections and infestations) | 1 (1)
Poly-contusion due to fall (Musculoskeletal and connective tissue disorders) | 1 (1)
Vomit (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Genital Herpes Virus infection (Infections and infestations) | 1 (1)
SARS-CoV-2 (Infections and infestations) | 1 (1)
Renal colic (Renal and urinary disorders) | 2 (2)
Leg ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Right conjunctival effusion (Eye disorders) | 1 (1)
Chlamydia trachomatis infection (Infections and infestations) | 1 (1)
Right eye hyposphagsma (Eye disorders) | 1 (1)
Lithotripsy (Hepatobiliary disorders) | 1 (1)
tympanic perforation (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT04097925/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT04097925/SAP_002.pdf
  • Informed Consent Form (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/25/NCT04097925/ICF_003.pdf